CLINICAL TRIAL: NCT03933085
Title: Spanish Translation and Cultural Adaptation of the Memory Support System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Octavio A. Santos, Prinicpal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-008125
Record Dates: First submitted 2019-03-13; First posted 2019-05-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Mild Cognitive Impairment
Keywords: Spanish-Speaking; Hispanic; ages ≥50
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MCI Group (Experimental): A within-subject, multiple baseline design, with each subject serving as their own control,4 will be implemented to get the maximum number of participants trained in the use of the MSS during the proposed funding period. This 2-year study will involve four phases: a 4-month translation and cultural adaptation development phase, a 12-month recruitment and treatment implementation phase, a 6-month post data collection only phase, and a 2-month data analysis and result writing phase. Data analyses will be conducted using the Statistical Package for the Social Sciences (SPSS) program.
  Interventions: Behavioral: Memory Support System (MSS)

INTERVENTIONS:
Behavioral: Memory Support System (MSS) — A calendar/notetaking system focused on training a person with MCI to use a specific external memory compensatory strategy to complete relevant IADLs independently.

SUMMARY:
This study seeks to translate a proven cognitive treatment for Spanish-speaking Hispanics with subjective memory/cognitive complaints or a diagnosis of mild cognitive impairment (MCI) and their care partners. MCI causes cognitive changes that are noticed by the individual or others. These changes do not significantly interfere with independence. MCI also increases the risk of developing Alzheimer's or another dementia, particularly in Hispanics/Latinos. There is no medication that improves cognition or delays MCI. However, providing cognitive treatment can alleviate the effects of MCI. Only a few cognitive interventions have been proven effective in the U.S., but none has been adapted to the Spanish-speaking Hispanic community. Our proposed cognitive treatment uses effective strategies (e.g., calendar and notetaking) to compensate for memory loss. The investigators will first follow international guidelines to ensure proper translation of our treatment into Spanish. Then, the investigators will pilot test our translated intervention in 20 Spanish-speaking Hispanic participants with subjective memory/cognitive complaints or a diagnosis of MCI and their care partners (40 participants total). The investigators will also assess the degree to which participants follow medical advice; their beliefs in their ability to succeed in and do daily activities, including managing medications; their feelings and potential burden associated with caregiving before and after the treatment as well as 8 weeks later. Results will allow the investigators to determine whether our treatment was effective and to calculate the number of participants required for larger studies. Overall, the study represents an important step to respond to the needs of the Hispanic community.

DETAILED DESCRIPTION:
Mild cognitive impairment (MCI) constitutes a high-risk state for conversion to dementia, making the search for interventions an urgent priority. In the absence of medications or dietary agents that improve cognition or delay MCI progression, offering nonpharmacological care approaches is currently considered good practice. Despite that, there are only a few evidence-based cognitive interventions for individuals with MCI available in the U.S. and, to the best of our knowledge, none is culturally sensitive to Hispanics; a group more prone to Alzheimer's disease or other dementias compared to non-Hispanic Whites. The overall goal and primary aim of this pilot project is to translate and begin to culturally adapt an evidence-based compensatory cognitive rehabilitation intervention, the Memory Support System (MSS), for Spanish-speaking Hispanics with subjective memory/cognitive complaints or a diagnosis of MCI and their care partners residing in the U.S. The MSS is a calendar/notetaking intervention proven effective in helping those with MCI compensate for memory loss in day-to-day function. Translation of the MSS and other materials will follow international guidelines. The Spanish MSS will be piloted in a sample of 20 participants in a within-subject, pre- and post-intervention assessment design. Outcome measures of program adherence, functional memory/general ability, self-efficacy, mood, anxiety, medication management skills, quality of life, and caregiver burden will be administered before and after the intervention, as well as at 8-week post-intervention to estimate effect size for power analyses for use in a future between-subject random assignment multicenter clinical trial. Overall, this pilot project represents an important step to significantly contribute to the development and promotion of clinical neuropsychological interventions responsive to the needs of the Hispanic community.

ELIGIBILITY:
Inclusion Criteria:

* Subjective memory/cognitive complaints or a diagnosis of single or multi-domain MCI
* Global score of ≤0.5 on the Clinical Dementia Rating (CDR)
* Scores of ≥4 on items six to nine on the Linguistic History Form (CLS) and scores of ≤6 on items on the Functional Assessment Scale (FAS), when applicable, from the Spanish language Uniformed Data Set (UDS) from the National Alzheimer's Coordinating Center's (NACC);
* A score of ≥115 on the Spanish Translation of the Dementia Rating Scale-Second edition (ST-DRS-2);
* Having contact with a cognitively normal care partner screened with the Mini Mental Status Examination (MMSE ≥24) at least twice a week; and
* Either not taking or stable on nootropic(s) for at least 3 months.

Exclusion Criteria:

* Visual/hearing impairment and/or history of reading or written inability/disability sufficient to interfere with MSS training; and/or
* Inclusion in another clinical trial that would exclude participation; subject will be considered for participation at the end of such a trial or as appropriate.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Memory Support System (MSS) adherence at 2 weeks after intervention start and at 2-month follow-up | 2 weeks after intervention start and 2-month follow-up
  To assess MSS adherence (i.e., how well a participant with subjective memory/cognitive complaints or a diagnosis of MCI utilizes all the MSS sections), the therapist will rate each participant based upon four criteria (≥7/10 scores considered compliant) for 2 days randomly selected.

SECONDARY OUTCOMES:
Change from Baseline Memory functional ability at 2 weeks after intervention start and at 2-month follow-up | 2 weeks after intervention start and 2-month follow-up
  To assess memory functional ability, care partners will complete a modified version of the Memory Subscale of the Everyday Cognition (E-Cog) at all assessment points. The E-Cog scores range from 8 to 32, where lower scores represent better memory functional ability.
Change from Baseline Self-efficacy at 2 weeks after intervention start and at 2-month follow-up | 2 weeks after intervention start and 2-month follow-up
  To assess self-efficacy, participants with subjective memory/cognitive complaints or a diagnosis of MCI will complete a modified version of specific subscales the Self-Efficacy in Memory scale (SEM) (Do Chores, Social/Recreational Activities, and Manage Disease in General) of the Chronic Disease Self-Efficacy Scales at all assessment points. The SEM scores range from 9 to 90, where higher scores represent better self-efficacy.
Change from Baseline Mood at 2 weeks after intervention start and at 2-month follow-up | 2 weeks after intervention start and 2-month follow-up
  To assess mood, participants with subjective memory/cognitive complaints or a diagnosis of MCI and care partners will complete the Center for Epidemiological Studies Depression Scale (CES-D) at all assessment points. The CES-D scores range from 0-60, where higher scores represent more symptoms of depression.
Change from Baseline Anxiety at 2 weeks after intervention start and at 2-month follow-up | 2 weeks after intervention start and 2-month follow-up
  To assess anxiety, participants with subjective memory/cognitive complaints or a diagnosis of MCI and care partners will complete the Anxiety Inventory Form from the State-Trait Anxiety Inventory by the Resources for Enhancing Alzheimer's Caregiver Health project (REACH) at all assessment points. The REACH scores range from 10-40, where higher scores represent more symptoms of anxiety.
Change from Baseline Quality of Life at 2 weeks after intervention start and at 2-month follow-up | 2 weeks after intervention start and 2-month follow-up
  To assess quality of life, participants with subjective memory/cognitive complaints or a diagnosis of MCI and care partners will complete the Quality of Life in Alzheimer's Disease measure (QoL-AD) at all assessment points. The QoL-AD scores range from 13-52, where higher scores represent better quality of life.
Change from Baseline General Functional Ability at 2 weeks after intervention start and at 2-month follow-up | 2 weeks after intervention start and 2-month follow-up
  To assess general functional ability, care partners will complete the Functional Assessment Scale (FAS)
Change from Baseline Caregiver Burden at 2 weeks after intervention start and at 2-month follow-up | 2 weeks after intervention start and 2-month follow-up
  To assess caregiver burden, care partners will complete the Caregiver Burden Interview-Short Form (CBI-SF) at all assessment points. The CBI-SF scores range from 0-48, where higher scores represent more care giver burden.
Change from Baseline Medication Management Skills at 2 weeks after intervention start and at 2-month follow-up | 2 weeks after intervention start and 2-month follow-up
  To assess medication management skills, participants with subjective memory/cognitive complaints or a diagnosis of MCI will complete the Pillbox Test (PT) at all assessment points (≥5 errors considered failure).

OTHER OUTCOMES:
Intervention evaluation by participants and support partners | 2-month follow-up
  To evaluate intervention at the end of MSS training, each dyad will undergo a qualitative semi-structured interview by the therapist about the training process itself, seeking suggestions for improving the MSS, teaching curriculum, and intervention logistics.

CONTACTS AND LOCATIONS:
Overall Officials: Octavio A Santos, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
All published reports will be of a summary nature, and no individual research subjects will be identified except to the investigative staff involved and only for research purposes. No personal identifying data will be released on subjects without prior consent from the subject. Data will be obtained from study participants via clinical records and interaction with the principal investigator (PI) (Dr. Santos) and/or PI's supervisors (Drs. Chandler and Pedraza). The proposed study will utilize webbased electronic data capture forms using Research Electronic Data Capture (REDCap) software previously created for use in other studies and stored on a server hosted by the Mayo Clinic Center for Translational Science Activities (CTSA) (Grant UL1 RR024150). REDCap is a secure Web-based application for building and managing online databases for clinical research studies. Information in REDCap will be scrubbed of Protected Health Information and utilize research IDs.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials